CLINICAL TRIAL: NCT02896764
Title: Interest of the Cone-beam Computed Tomography in the Imagery of the Middle Ear
Acronym: ECCO1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MWS_2014_14
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Ear Diseases
MeSH Terms: conditions — Ear Diseases | interventions — Cone-Beam Computed Tomography

ARMS (1):
- Eligible patients for cone-beam CT (Experimental): A cone-beam CT will be offered to the patient undergoing a CT scan of the middle ear
  Interventions: Device: Cone-beam CT

INTERVENTIONS:
Device: Cone-beam CT

SUMMARY:
Cone beam computed tomography (CBCT), is a recent medical imaging technique where the X-rays are divergent, forming a cone.

As a result, this technique is less irradiating that the scanner. The purpose of this exploratory study is to compare the performance of the scanner and the cone beam in the detection of anatomical structures of the ear.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Indication of a CT scan of the ear
* Written and signed informed consent by the patient to participate in the study

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Patient under a legal protection procedure
* Lack of affiliation to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the cone-beam CT vs CT scan | 1 minute
  Correlation coefficient measuring the concordance for a given radiologist, between the number of anatomical structures of the ear viewed by the cone beam CT and the CT scanner on a total of 24 studied structures

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A de Rothschild, Paris, France